CLINICAL TRIAL: NCT04197752
Title: Use of Regional Anesthesia and Analgesia Techniques in Obese Patients: A Prospective Observational Study
Brief Title: Regional Anesthesia and Analgesia Techniques in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emine Aysu Salviz, MD, Associate Professor, Istanbul University
Other Study IDs: 2019/664
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Regional Anesthesia
Keywords: Obesity; Neuroaxial blocks; Peripheral nerve blocks; Performance; Complication
MeSH Terms: conditions — Obesity | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients: Body mass index > 30 kg/m2
  Interventions: Other: Regional anesthesia/analgesia techniques
- Non-obese patients: Body mass index < 30 kg/m2
  Interventions: Other: Regional anesthesia/analgesia techniques

INTERVENTIONS:
Other: Regional anesthesia/analgesia techniques — Neuroaxial or peripheral block anesthesia/analgesia technique that is appropriate for the patient's surgery

SUMMARY:
Obesity is a health problem throughout the world and has increasingly become a widespread epidemic all over the world and also in Turkey. Anesthesia management of obese patients is challenging because of difficult airway, increased drug doses, co-morbidities, loss of anatomical landmarks and difficulties in positioning.

Neuroaxial and peripheral nerve blocks are widely used in anesthesia practice in both obese and non-obese patients undergoing different surgical operations.

In this prospective observational study, the investigators plan to enroll all patients that are applied neuroaxial or peripheral blocks during the study period. The aim of this study is to compare the differences and difficulties of regional anesthesia/analgesia techniques in obese and non-obese patients.

DETAILED DESCRIPTION:
Obesity is a health problem throughout the world and has increasingly become a widespread epidemic all over the world and also in Turkey. Anesthesia management of obese patients is challenging because of difficult airway, increased drug doses, co-morbidities, loss of anatomical landmarks and difficulties in positioning.

On the other hand, neuroaxial and peripheral nerve blocks are widely used in anesthesia practice in both obese and non-obese patients undergoing different surgical operations.

In this prospective observational study, the investigators plan to enroll all patients that are applied neuroaxial or peripheral blocks during the study period. The difficulty of block performance, its relationship with experience, the requirement of changing hands with more experienced clinician, the requirement of changing patient position, regional anesthesia approach or needle (size and length), the requirement of adding rescue block, block success, performance duration, the number of needle direction (multiple attempts), the requirement of changing anesthesia or analgesia technique (conversion to general anesthesia), the requirement of adding another block monitorisation technique, adverse effect/complication, patient satisfaction and patient's request for a similar technique next time are all recorded both in obese and non-obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for regional anesthesia/analgesia
* > 18 years old
* ASA 1-3

Exclusion Criteria:

* < 18 years old
* Patient refusal for regional anesthesia/analgesia
* Patient refusal to participate in the study
* Allergic to local anesthetics
* Psychiatric diseases
* Incapable to communicate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient eligible for regional anesthesia/analgesia procedures
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The difficulty of block performance | through the block performance, within 5-10 minutes
  0: easy, 1: difficult, 2: very difficult

SECONDARY OUTCOMES:
The experience of the anesthesiologist | through the Anesthesiology residency training period, within 5 years and Anesthesiology experience, within 20 years
  0: Junior resident, 1: senior resident, 2: attending anesthesiologist, 3: assoc.prof./prof.anesthesiologist
The requirement of changing hands with a more experienced anesthesiologist | through the block performance, within 5-10 minutes
  The number of changing
The requirement of changing patient position | through the block performance, within 5-10 minutes
  Yes/No
The requirement of changing regional anesthesia/analgesia approach | through the block performance, within 5-10 minutes
  Yes/No
The requirement of changing needle size or length | through the block performance, within 5-10 minutes
  Yes/No
The requirement of adding rescue block | through the block performance, within 5-10 minutes
  Yes/No
Block performance duration | 0-30 minutes
  Time period
The number of needle direction | through the block performance, within 5-10 minutes
  Number
The requirement of conversion to general anesthesia | through the block performance, within 5-10 minutes
  Yes/No
The requirement of adding another block monitorization technique | through the block performance, within 5-10 minutes
  Yes/No
Adverse effect/complication rate | 1 week
  Yes/No
Block success | 0-30 minutes
  Yes/No
Patient satisfaction | 1 week
  0-3 (0: not satisfied...3: very satisfied)
Patient's request for a similar technique next time | 1 week
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Emine A Salvız, M.D., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franco CD, Gloss FJ, Voronov G, Tyler SG, Stojiljkovic LS. Supraclavicular block in the obese population: an analysis of 2020 blocks. Anesth Analg. 2006 Apr;102(4):1252-4. doi: 10.1213/01.ane.0000198341.53062.a2. PMID 16551933
- [Background] Hanouz JL, Grandin W, Lesage A, Oriot G, Bonnieux D, Gerard JL. Multiple injection axillary brachial plexus block: influence of obesity on failure rate and incidence of acute complications. Anesth Analg. 2010 Jul;111(1):230-3. doi: 10.1213/ANE.0b013e3181dde023. Epub 2010 Apr 24. PMID 20418535